CLINICAL TRIAL: NCT02797145
Title: Intensive Versus Conventional Digoxin Use in Patients With Heart Failure: a Randomized Controlled Trial
Brief Title: Intensive Versus Conventional Digoxin Use in Patients With Heart Failure
Acronym: ICHF
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Ana Nery (Other)
Responsible Party: Principal Investigator, Andre Duraes, PhD, Coordinator, Hospital Ana Nery
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 52553116.7.0000.0045
Record Dates: First submitted 2016-05-26; First posted 2016-06-13 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-06

CONDITIONS: Heart Failure
Keywords: Digoxin
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive Group (Active Comparator): Dose adjusted digoxin by the recommended range for the serum digoxin: 0.5-0.9 nanogram/mL
  Interventions: Drug: Digoxin dose-adjusted
- Conventional (Placebo Comparator): Use digoxin as recommended by the guidelines.
  Interventions: Drug: Standard dose

INTERVENTIONS:
Drug: Digoxin dose-adjusted — Serum digoxin concentration : 0.5 to 0.9 nanogram/mL
  Other Names: Intensive Digoxin
  Arms: Intensive Group
Drug: Standard dose — the dose of digoxin will be determined at the physician's discretion using traditional dosing methods.
  Other Names: Conventional dose
  Arms: Conventional

SUMMARY:
Digoxin was approved for heart failure treatment in 1998 according to current regulations made by Food and Drug Administration (FDA), based on the following clinical trials: The Prospective and Randomized Study of Ventricular Function and Efficacy of Digoxin (PROVED), Randomized Assessment of Digoxin on Inhibitors of the Angiotensin Converting Enzyme (RADIANCE) and Digitalis Investigation Group (DIG). Also, it was approved for the control of ventricular response rate in atrial fibrillation patients.

Several clinical trials with digoxin provided convincing evidence that support the digoxin use heart failure (HF) treatment of symptomatic patients. PROVED trial was a placebo-controlled, twelve weeks duration study. This study included patients with decreased systolic function, sinus rhythm and heart failure stable symptoms, these patients were using digoxin and diuretics. Patients whom digoxin was removed presented a twice heart failure worsen, reduction of exercise capacity and also a reduction of left ventricle ejection fraction, in comparison to patients that kept the digoxin therapy. The study RADIANCE followed a similar protocol; however the patients used ACE inhibitors besides digoxin and diuretics. The digoxin removal was associated with a six times worsen of heart failure, despite the maintenance of ACE inhibitors and diuretics. There was a worsening in the functional capacity, life quality and in the ejection fraction on the digoxin removal patients' group.

DETAILED DESCRIPTION:
The benefits of digoxin can be related not only with its hemodynamic effects, but also its capacity to improve the neuro hormonal profile. Improvements on the neurohormonal profile and on hemodynamic occur with low doses of digoxin, and the dose increment not always results in improving effects. In the studies PROVE e RADIANCE the clinical benefits were similar among patients with low digoxin serum (serum < 1ng/mL) and those with high dose of digoxin serum. One current post-hoc analysis of DIG study, that included patients with preserved systolic function or reduced systolic function, suggested a survival benefit for the patients with < 1,0 ng/mL digoxin serum.

Several studies documented the effectiveness of digoxin to reduce clinically relevant outcomes in HF patients. These studies showed symptomatic improvement of aerobic capacity and life quality in patients with symptomatic HF (functional class II-IV). Such benefits occur independently of basal rhythm or HF aetiology. It is important to highlight that these studies were performed in a period before the BB utilization in the systolic HF treatment. On the other hand, on side of DIG study evaluate the digoxin effect versus placebo in patients with preserved eject. The use of digoxin has no effect in the mortality or in the hospitalization due to cardiovascular causes. There was a tendency to reduce the hospitalization due to HF worsening; however there was also an increase tendency of increase hospitalization due to unstable angina. Currently was documented that digoxin serum levels above 1,0 ng/dL are associated with high chance of death, in retrospective analysis of SOLVD and DIG studies. The subgroup that kept the digoxin serum levels between 0,3 and 0,9 ng/mL had the greater benefit, including less mortality between men. From these findings, it began recommending low doses of digoxin in order to get this serum levels. Remains the discussion if the utilization of serum levels as therapeutic guidelines bring any additional benefit. The PROVED and RADIANCE studies showed the necessity to keep the digoxin use in symptomatic HF patients, otherwise functional class worsening and increase of hospitalization chance.[2] However, the long-term effect of digoxin on mortality and hospitalization for heart failure or other causes is unknown. The use of digoxin increases the intracellular concentration of calcium ions, increasing the platelet activation and favoring the occurrence of thromboembolic events. This fact is particularly dangerous because patients with AF have increased susceptibility to suffer ischemic stroke due to thromboembolic events. Besides, high numbers of drugs used in the management of patients with HF reduces renal clearance and supports the elevation of serum digoxin concentration and increased toxicity and mortality by arrhythmias. (OUYANG et al., 2015) (WHITBECK et al., 2013).

It is worth noting that the DIG study excluded from trial patients with AF, and has carried out strict control of digoxin serum levels. These two facts taken together may have collaborated with digoxin action of neutrality on mortality rates. A particular concern is the fact that elevated digoxin serum levels have been correlated with increased mortality in multiple patient populations. The AFFIRM study identified association of digoxin use with all-cause mortality (1.41, 95% CI 1.19-1.67, P<0.001); cardiovascular mortality (1.35, 95% CI 1.06-1.71, P<0.016); and deaths from arrhythmias (1.61, 95% CI 1,12-2,30, P<0,009)(WHITBECK et al., 2013). By contrast, the AFFIRM study did not held control of digoxin serum levels of patients using digoxin. The RIKS-HIA study evaluated outcome after 1 year in 4426 patients with AF and without congestive heart failure using digoxin, and identified increased overall mortality with a relative risk estimated at 1.42 (95% CI 1.29 to 1 , 56%) when compared to 16,587 control patients. Another study that was performed to investigate better the effects of digoxin was the TREAT-AF (The Retrospective Evaluation and Assessment of Therapies in AF) study. This study was a retrospective cohort study of patients with newly diagnosed AF treated in the U.S. Department of Veterans Affairs (VA) healthcare system. The TREAT-AF compared data of patients treated with digoxin against patients non-treated with digoxin. The results showed that digoxin treatment was significantly associated with death in the multivariate Cox regression model (hazard ratio [HR]: 1.26, 95% confidence interval [CI]: 1.23 to 1.29, p < 0.001) and after propensity matching (HR: 1.21, 95% CI: 1.17 to 1.25, p < 0.001). Also the cumulative incidence of death was higher in the digoxin-treated patients versus the untreated group (p < 0.001). The TREST-AF outcomes exalted once again the need for further investigation about the digoxin effects. Observational data have generally come to similar conclusions. In a large study of 2,892 Kaiser patients with newly diagnosed heart failure with reduced ejection fraction (HFrEF), of whom 22.9% had AF, incident digoxin use was associated with higher mortality (HR: 1.72; 95% CI: 1,25 to 2.36), but there was no significant difference in the risk of HF hospitalization (HR: 1.05; 95% CI0.82 to 1.34). The ATRIA-CVRN (Anti-coagulation and Risk factors in Atrial Fibrillation-Cardiovascular Research Network) study, which was a propensity score matching analysis of 14,787 Kaiser patients with incident AF and without HF, found that incident digoxin use was independently associated with higher risk of death (HR: 1.71; 95% CI: 1.52 to 1.93) and a higher risk of hospitalization (HR: 1.63; 95% CI: 1.56 to 1.71). (ALLEN et al., 2015)

ELIGIBILITY:
Inclusion Criteria:

* Heart Failure with reduced EF (< 40%) and sinusal rhythm or atrial fibrillation

Exclusion Criteria:

* Pregnant women
* Any degree of atrioventricular block
* Renal failure (Creatinine Clearance lower than 50 mL/min)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-05; Primary Completion 2018-05 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with improvement in functional class and free of hospital admissions | one year
  Digoxin can still be useful in people who remain symptomatic despite proper diuretic and ACE inhibitor treatment.
Proportion of patients with adverse events: loss of appetite, nausea, vomiting, abdominal pain, diarrhea, blurred vision and or new atrial or ventricular extrasystoles. | one year
  Common adverse effects (≥1% of patients) include loss of appetite, nausea, vomiting, and diarrhea as gastrointestinal motility increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital ana Nery, Salvador, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: Undecided